CLINICAL TRIAL: NCT05502913
Title: Fecal Microbiota Transplantation to Improve Efficacy of Immune Checkpoint Inhibitors in Metastatic Lung Cancer
Brief Title: Fecal Microbiota Transplantation With Immune Checkpoint Inhibitors in Lung Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Soroka University Medical Center (Other)
Collaborators: Biotax Labs LTD (Industry); Israel Cancer Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: sor 0173-21 ctil
Record Dates: First submitted 2022-08-08; First posted 2022-08-16 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Metastatic Lung Cancer
Keywords: Fecal microbiome transplant; Metastatic lung cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Anti-Bacterial Agents; Rifaximin; Fecal Microbiota Transplantation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard of care (SoC) (IO±CTX) + FMT (Experimental): Subjects assigned to Arm 1 will be required to swallow FMT capsules in a regimen of ten capsules in the morning and ten capsules in the afternoon on day 1 of the first (chemo-)immunotherapy cycle, and then every three weeks.
  abbreviation: Immuno-Oncology (IO) Chemotherapy (CTX)
  Interventions: Drug: Antibiotics; Other: FMT (Fecal Microbiota Transplantation)
- standard-of-care treatment (No Intervention): Subjects will receive standard-of-care treatment only.

INTERVENTIONS:
Drug: Antibiotics — Recipients will undergo bowel preconditioning with antibiotics (Rifaximin) following randomization.
  Other Names: Rifaximin
  Arms: standard of care (SoC) (IO±CTX) + FMT
Other: FMT (Fecal Microbiota Transplantation) — FMT involves the transplantation of fecal bacteria from a screened donor to a recipient. This will be achieved per os in the form of a capsule containing freeze-dried stool obtained from the donor.
  Arms: standard of care (SoC) (IO±CTX) + FMT

SUMMARY:
Immunotherapy has recently become a main-stream treatment option in cancer care, with improved clinical outcomes in many malignancies, especially that of lung cancer. The long-term benefits of this treatment however are limited. There is therefore a critical need to distinguish predictive biomarkers of response from those of resistance, and to develop synergistic strategies for improved therapeutic response. Strong emerging evidence indicates that the gut microbiome has the ability to influence response to immunotherapy. Unlike tumor genomics, the gut microbiome is modifiable, and thus its modulation to enhance response to immunotherapy is an attractive therapeutic strategy.

Working hypothesis: Fecal Microbiota Transplant (FMT) treatment in conjunction with standard (chemo-)immunotherapy as a first-line treatment for metastatic lung cancer enhances disease control rate.

The main objective of this study is to evaluate the safety and efficacy of Fecal Microbiota Transplant (FMT) in altering response to immunotherapy in patients with metastatic lung cancer. The overall goal is to determine microbiome compositional and gene-content changes in patients who respond more efficiently to immunotherapy subsequent to FMT. This understanding may lead to future microbiome-based treatments in combination with immunotherapy to significantly increase lung cancer treatment efficacy. In this prospective clinical and molecular study, we will perform an in-depth analysis of the potential role of FMT in the context of immunotherapy.

DETAILED DESCRIPTION:
Only a small subset of tumor types benefit from immune checkpoint inhibitor therapy, where most responders eventually develop resistance. Oral administration of Fecal Microbiota Transplantation (FMT) from treatment-responsive patients has been found to considerably improve Programmed death-ligand 1 (PD-L1)-based immunotherapy outcomes as well as inhibit tumor growth through augmented dendritic cell and T cell responses.

This study aims to investigate the safety and efficacy of FMT treatment combined with first-line (chemo-)immunotherapy in metastatic lung cancer. The study will include a thorough microbiome composition analysis of FMT donors and recipients to be correlated to clinical outcomes. In addition, blood samples will be analyzed using a novel commensal antigen microarray for rapid serum profiling.

Patients with metastatic malignancy who completely respond to immunotherapy will serve as the fecal implant donors. Dr. Arik Segal's Lab will produce capsules with one donor/capsule. In an open-label approach, patients will receive FMT on the first day of (chemo-)immunotherapy cycle one and every 3-4 weeks based on the specific (chemo-)immunotherapy protocol. Before FMT treatment, participants will receive active antibiotics. The second arm will receive standard-of-care treatment only. Study participants will be evaluated throughout the study using imaging, laboratory, vital signs, and disease status assessments until the end of the study.

Stool samples from study participants will be collected before the start of treatment during the (chemo-)immunotherapy cycle and at the end of treatment for sequencing and bioinformatics analysis of the microbiome. Blood samples will be collected from all donors at the study start and from all recipients at recruitment, on the day of each FMT administration, and at the end of treatment.

Statistics:

A one-sided test for differences in proportions and type I error of 0.05 will have a power of 88% to detect a 30% difference in response between the FMT and placebo group, for a total of 80 randomized patients, 40 in each treatment group stratified by PD-L1 status.

ELIGIBILITY:
Patient (Recipient) Inclusion Criteria:

1. A histologically confirmed diagnosis of malignancy.
2. Patients over the age of 18.
3. Patients planning to be treated with chemotherapy, immune checkpoint inhibitors and/or targeted therapy.
4. Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2
5. Able to provide written informed consent.

Patient (Recipient) Exclusion Criteria:

1. Severe or life-threatening food allergy (e.g. nuts, seafood)
2. Allergy or other contraindication to omeprazole, investigational medicinal product.
3. Treatment with pre- or probiotics in the four weeks prior to randomization.
4. Severe immunodeficiency:

   * Systemic chemotherapy <30 days from baseline
   * Known neutropenia with absolute neutrophils <1.0x109 cells/µL
   * Prolonged treatment with corticosteroids (equivalent to prednisone >60mg daily for >30 days) within 8 weeks of randomization
5. Swallowing disorder, oral-motor discoordination, inability to swallow capsules
6. Pregnant or breastfeeding or expecting to conceive or father children within the trial's projected duration, starting from the pre-screening or screening visit through to 120 days after the last dose of trial treatment.

Donor Inclusion Criteria:

1. A histologically confirmed diagnosis of malignancy.
2. Over the age of 18.
3. Treated with immune checkpoint inhibitors and with a full response.
4. Currently attending medical follow-ups

Donor Exclusion Criteria:

1. Has not consumed any antimicrobials within the past 3 months
2. No prior exposure to HIV or viral hepatitis or suffering from tuberculosis/latent tuberculosis
3. No risk factors for blood-borne viruses, including high-risk sexual behavior, use of illicit drugs, any tattoo/body piercing/needlestick injury/blood transfusion/acupuncture, all within the past 6 months
4. No signs or symptoms consistent with Coronavirus disease 19 (COVID-19) or a nose/throat and/or stool sample with detectable Coronavirus disease 2 (CoV-2)
5. Has not received a live attenuated vaccine within the past 6 months
6. No underlying gastrointestinal conditions/symptoms (e.g., history of IBD, irritable bowel syndrome (IBS), chronic diarrhea, chronic constipation, coeliac disease, bowel resection or bariatric surgery)
7. No acute diarrhea/gastrointestinal symptoms within the 2 weeks prior to donating
8. No family history of any significant gastrointestinal conditions (e.g., family history of inflammatory bowel disease (IBD) or colorectal cancer)
9. No history of atopy (e.g., asthma, eosinophilic disorders)
10. Does not suffer from any systemic autoimmune conditions
11. Does not start any new treatment regimens within 2 weeks of fecal collection
12. No neurological or psychiatric conditions or known risk for prion disease
13. No history of chronic pain syndromes, including chronic fatigue syndrome and fibromyalgia
14. No history of receiving growth hormone, insulin from cows or clotting factor concentrates
15. Has not received an experimental drug or vaccine within the past 6 months
16. No history of travel to tropical countries within the past 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) | up to 2 years
  PFS is defined as the time passed from screening until the date of progressive disease (PD) or death from any cause. Imaging will be performed using computed tomography (CT) and/or Positron emission tomography (PET).

SECONDARY OUTCOMES:
Overall Survival (OS) | up to 4 years
  OS is defined as the time passed from randomization until death from any cause.
Objective response rate (ORR) | From randomization (Day 0) until end of study
  ORR is defined as the percentage of subjects who had a complete response (CR) or partial response (PR), as defined by ir-RECIST v1.1, and is based on the best response obtained.
Rate of Disease Control | up to 2 years
  Rate of Disease Control is defined as the percentage of subjects who had a complete response (CR), partial response (PR), or stable disease (SD), as defined by ir-RECIST v1.1.
Microbiome analysis | up to 2 years
  Microbiome analysis of the stool of donors and recipients (before and after FMT) to reveal the optimum microbiome-based components to significantly increase cancer immunotherapy efficacy
Serum antibody levels and lymphocyte subpopulation distribution | up to 2 years
  Analysis of serum antibodies and blood lymphocyte repertoires to be correlated to gut microbes and yeasts via blood samples of donors and recipients at several timepoints prior and post FMT induction
Safety and feasibility | up to 2 years
  Number of adverse events and serious adverse events related definitely to fecal microbiota transplantation (FMT).

CONTACTS AND LOCATIONS:
Overall Officials: Ismaell Massalha, MD, Principal Investigator — Soroka University Medical Center
Locations (2):
- Israel (2):
  - Soroka Medical Center, Beersheba
  - Rabin Medical Center, Petah Tikva

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Robert C. A decade of immune-checkpoint inhibitors in cancer therapy. Nat Commun. 2020 Jul 30;11(1):3801. doi: 10.1038/s41467-020-17670-y. PMID 32732879
- [Background] Chen D, Wu J, Jin D, Wang B, Cao H. Fecal microbiota transplantation in cancer management: Current status and perspectives. Int J Cancer. 2019 Oct 15;145(8):2021-2031. doi: 10.1002/ijc.32003. Epub 2018 Dec 30. PMID 30458058
- [Background] Davar D, Dzutsev AK, McCulloch JA, Rodrigues RR, Chauvin JM, Morrison RM, Deblasio RN, Menna C, Ding Q, Pagliano O, Zidi B, Zhang S, Badger JH, Vetizou M, Cole AM, Fernandes MR, Prescott S, Costa RGF, Balaji AK, Morgun A, Vujkovic-Cvijin I, Wang H, Borhani AA, Schwartz MB, Dubner HM, Ernst SJ, Rose A, Najjar YG, Belkaid Y, Kirkwood JM, Trinchieri G, Zarour HM. Fecal microbiota transplant overcomes resistance to anti-PD-1 therapy in melanoma patients. Science. 2021 Feb 5;371(6529):595-602. doi: 10.1126/science.abf3363. PMID 33542131
- [Background] Baruch EN, Youngster I, Ben-Betzalel G, Ortenberg R, Lahat A, Katz L, Adler K, Dick-Necula D, Raskin S, Bloch N, Rotin D, Anafi L, Avivi C, Melnichenko J, Steinberg-Silman Y, Mamtani R, Harati H, Asher N, Shapira-Frommer R, Brosh-Nissimov T, Eshet Y, Ben-Simon S, Ziv O, Khan MAW, Amit M, Ajami NJ, Barshack I, Schachter J, Wargo JA, Koren O, Markel G, Boursi B. Fecal microbiota transplant promotes response in immunotherapy-refractory melanoma patients. Science. 2021 Feb 5;371(6529):602-609. doi: 10.1126/science.abb5920. Epub 2020 Dec 10. PMID 33303685
- [Background] Gopalakrishnan V, Spencer CN, Nezi L, Reuben A, Andrews MC, Karpinets TV, Prieto PA, Vicente D, Hoffman K, Wei SC, Cogdill AP, Zhao L, Hudgens CW, Hutchinson DS, Manzo T, Petaccia de Macedo M, Cotechini T, Kumar T, Chen WS, Reddy SM, Szczepaniak Sloane R, Galloway-Pena J, Jiang H, Chen PL, Shpall EJ, Rezvani K, Alousi AM, Chemaly RF, Shelburne S, Vence LM, Okhuysen PC, Jensen VB, Swennes AG, McAllister F, Marcelo Riquelme Sanchez E, Zhang Y, Le Chatelier E, Zitvogel L, Pons N, Austin-Breneman JL, Haydu LE, Burton EM, Gardner JM, Sirmans E, Hu J, Lazar AJ, Tsujikawa T, Diab A, Tawbi H, Glitza IC, Hwu WJ, Patel SP, Woodman SE, Amaria RN, Davies MA, Gershenwald JE, Hwu P, Lee JE, Zhang J, Coussens LM, Cooper ZA, Futreal PA, Daniel CR, Ajami NJ, Petrosino JF, Tetzlaff MT, Sharma P, Allison JP, Jenq RR, Wargo JA. Gut microbiome modulates response to anti-PD-1 immunotherapy in melanoma patients. Science. 2018 Jan 5;359(6371):97-103. doi: 10.1126/science.aan4236. Epub 2017 Nov 2. PMID 29097493